CLINICAL TRIAL: NCT00161785
Title: Investigation of the Seropersistence of TBE Antibodies and the Booster Response to FSME-IMMUN 0.5 ml in Adults Aged 18 - 67 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 223
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Tick-borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: FSME-IMMUN 0.5ml

SUMMARY:
The purpose of this study is to assess:

* TBE antibody persistence 2 and 3 years after the third TBE vaccination with FSME-IMMUN 0.5ml by means of ELISA and neutralization test (NT).
* TBE antibody response to a booster vaccination with FSME-IMMUN 0.5ml, by means of ELISA and NT.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects will be eligible for participation in this study if:

* they understand the nature of the study, agree to its provisions and provide written informed consent;
* they received the third vaccination with FSME-IMMUN 0.5ml during the course of Baxter Study 213;
* blood was drawn before and after their third vaccination during the course of Baxter Study 213;
* they showed an ELISA-concentration > 126 VIE U/ml and / or a NT-titer >= 1:10 after the third vaccination in Baxter Study 213;
* they agree to keep a Subject Diary.

Exclusion Criteria:

Subjects will be excluded from participation in this study if they:

* received any TBE vaccination since their third vaccination with FSME-IMMUN 0.5ml;
* received a vaccination against yellow fever and / or Japanese B-encephalitis since their third vaccination with FSME-IMMUN 0.5ml;
* are known to be HIV positive (a special HIV test is not required for the purpose of the study) since their third vaccination with FSME-IMMUN 0.5ml;
* have a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent level of other alcoholic beverages);
* have received a blood transfusion or immunoglobulins within one month to the first and second blood draw;
* have participated in another Baxter vaccine study within the last six months (with the exception of follow-up studies).

Subjects will not be eligible for booster vaccination if:

* they do not meet the inclusion/exclusion criteria;
* they are not clinically healthy, (i.e. the physician would have reservations vaccinating with FSME-IMMUN 0.5ml outside the scope of a clinical trial);
* they suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids) that can be expected to influence immunological functions;
* they have donated blood or plasma within one month to the booster vaccination;
* female of childbearing potential are pregnant or breastfeeding before the booster vaccination (positive pregnancy test result at the medical examination before the booster vaccination);
* they have shown an allergic reaction to one of the components of the vaccine since their third vaccination in Baxter Study 213;
* they are simultaneously participating in another clinical trial including administration of an investigational product within six weeks prior to the booster vaccination until the end of the study.

Subjects who meet the inclusion/exclusion criteria, but have a febrile illness (body temperature >= 38.0°C, measured orally) at the scheduled time of vaccination, will not be vaccinated until their body temperature returns to normal.

Subjects who have received any vaccination within two weeks prior to the booster vaccination will not be vaccinated until an interval of two weeks has passed.

If subjects have received antipyretics within 4 hours prior to the intended TBE vaccination, the vaccination should be performed at a later time.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340
Dates: Start 2004-06; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Konior, MD, Principal Investigator — Szpital Jana Pawla II Oddzial Neuroinfekcji, Krakow, Poland
Locations (2):
- Poland (2):
  - Hospital in Debica - Zespo Opieki Zdrowotnej w Debicy, Dębica
  - Szpital Jana Pawla II Oddzial Neuroinfekcji, Krakow